CLINICAL TRIAL: NCT05732727
Title: Intensification of Blood Pressure Lowering Therapeutics Based on Diuretics Versus Usual Management for Uncontrolled Hypertension IN Patients With Moderate to Severe Chronic Kidney Disease: an Open Label, a Cluster Randomized Controlled, Phase 3 Trial
Brief Title: Intensification of Blood Pressure Lowering Therapeutics Based on Diuretics Versus Usual Management for Uncontrolled Hypertension IN Patients With Moderate to Severe Chronic Kidney Disease
Acronym: THINK
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DR210320; 2022-501494-39-00 (Other: EU CT)
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Chronic Kidney Disease(CKD); Uncontrolled Hypertension
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled
Masking Description: The very nature of the intervention assessed prevents any form of blinding, neither for care providers, nor for patients.
  However, the primary outcome is a composite outcome of events which we plan to adjudicate. As a consequence, the primary outcome will be blindly assessed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Antihypertensive algorithm based on diuretics agents : the clinicians will adjust the drug therapy according to the antihypertensive algorithm based on diuretics agents.
  Interventions: Drug: Antihypertensive algorithm
- Control group (Active Comparator): Standard of care : the clinicians will adapt the antihypertensive strategy according to his own standard of care which can be pharmacological or non-pharmacological therapies.
  Interventions: Drug: Standard of care

INTERVENTIONS:
Drug: Antihypertensive algorithm — Antihypertensive algorithm based on diuretics agents
  Arms: Experimental group
Drug: Standard of care — standard of care management for antihypertensive therapy intensification
  Arms: Control group

SUMMARY:
Chronic kidney disease (CKD) is a major public health issue worldwide. Hypertension is the first risk factor in patients with CKD for mortality, cardiovascular disease and end-stage renal disease. It's now well established that lowering blood pressure (BP) reduces renal and cardiovascular complications in this high-risk population. In the general population, in addition to lifestyle interventions, the strategy to initiate and escalate a BP-lowering drug treatment is well described. The drug therapies recommended to achieve optimal BP control in the general population are the following: blockers of the renin-angiotensin system (angiotensin-converting enzyme inhibitors (ACEi) or angiotensin receptor blockers (ARB)), diuretics (thiazides and thiazide-like diuretics), and calcium channel blockers. For patients with CKD, the guidelines advise to start the BP-lowering agent with ACEi or ARB, but then, there is no strong evidence to support the preferential use of any particular agent in controlling BP and the results of clinical trials are discordant. In the NephroTest cohort, a French cohort of patients with CKD stage 1 to 5, among 2015 patients, 1782 had hypertension, only 54% had a diuretic and 44% had uncontrolled hypertension. In this cohort, extracellular fluid (ECF) overload was an independent determinant of hypertension, uncontrolled hypertension and apparent treatment resistant hypertension. In the same cohort, ECF overload was independently associated with end-stage kidney disease and death. Our hypothesis is that patients with CKD and uncontrolled hypertension are fluid overloaded and that the second line of treatment after an ACEi or an ARB should be a diuretic. We hypothesize that a specific algorithm to lower BP in patients with moderate to severe CKD based on diuretics will be more effective in term of cardiovascular event, mortality and evolution to end-stage kidney disease as compared to standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Male or female >=18 years with a clinical frailty score ≤5 for patient aged over 80
* Advanced or moderate chronic kidney disease (eGFR 15 to 44.9 mL/min/1.73m² using CKD-EPI formula)
* Arterial hypertension treated with at least one blood pressure lowering drug therapy among blockers of the renin-angiotensin system (ACEi or ARB), at the maximal posology tolerated by the patients stable since at least one month. Other blood pressure lowering drug therapies are tolerated in combination with or in the event of intolerance to ACE inhibitors or ARBs.
* Uncontrolled office BP
* Uncontrolled office BP (>140 and/or 90 mmHg) confirmed by home blood pressure monitoring (>135 and/or 85 mmHg) or Day-time Ambulatory Blood Pressure Monitoring
* Participant covered by or entitled to social security
* Written informed consent obtained from the participant

Exclusion Criteria:

* Patient following any measures of legal presentation
* Pregnant or breastfeeding woman
* woman of childbearing without a highly effective contraceptive measure (combined or progestogen-only hormonal contraception associated with inhibition of ovulation, intrauterine device or intrauterine hormone-releasing system)
* Clinical signs of hypovolemia
* Symptomatic orthostatic hypotension
* Hyponatremia (<130 mmol/L)
* Dyskalemia (<3,5 mmol/L or >5,5 mmol/L)
* Major adverse cardiovascular event during the last three months: myocardial infarction, heart failure hospitalization, stroke
* Current medical history of cancer requiring chemotherapy
* Solid organ transplantation
* Two or more diuretic agents (loop diuretic, thiazides and thiazide-like diuretics)
* Mineralocorticoid receptor antagonists
* Autosomal dominant polycystic kidney disease treated with Tolvaptan
* Contraindication to diuretics involved in the algorithm
* Severe heart failure (NYHA III_IV)
* Cirrhosis Child B-C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
End stage kidney disease | Up to 36 months
  The primary endpoint is a time to event outcome, considering the following composite endpoint:
  * End stage kidney disease
  * eGFR decline of at least 40%
  * Cardiovascular events among myocardial infarction, heart failure, hospitalization and stroke
  * All cause mortality
eGFR decline of at least 40% | Up to 36 months
  The primary endpoint is a time to event outcome, considering the following composite endpoint:
  * End stage kidney disease
  * eGFR decline of at least 40%
  * Cardiovascular events among myocardial infarction, heart failure, hospitalization and stroke
  * All cause mortality
Cardiovascular events | Up to 36 months
  The primary endpoint is a time to event outcome, considering the following composite endpoint:
  * End stage kidney disease
  * eGFR decline of at least 40%
  * Cardiovascular events among myocardial infarction, heart failure, hospitalization and stroke
  * All cause mortality
All cause mortality | Up to 36 months
  The primary endpoint is a time to event outcome, considering the following composite endpoint:
  * End stage kidney disease
  * eGFR decline of at least 40%
  * Cardiovascular events among myocardial infarction, heart failure, hospitalization and stroke
  * All cause mortality

SECONDARY OUTCOMES:
Time to end-stage kidney disease | Up to 36 months
  All components of the composite endpoint will be assessed separately
Time to eGFR decrease of at leat 40% | Up to 36 months
  All components of the composite endpoint will be assessed separately
Time to the first cardiovascular event among myocardial infarction, heart failure, hospitalization and stroke | Up to 36 months
  All components of the composite endpoint will be assessed separately
All-cause mortality | Up to 36 months
  All components of the composite endpoint will be assessed separately
Change from baseline in blood pressure | From baseline and up to 36 months
  Systolic and diastolic blood pressure at months 3 and 6 then every 6 months (home blood pressure monitoring and office blood pressure measurement),
Proportion of patients with controlled blood pressure | 24 months
  Proportion of patients with controlled blood pressure at 2 years (PA< 135/85mmHg with home blood pressure monitoring)
Change from baseline in glomerular filtration rate | From baseline and up to 36 months
  Change from baseline in glomerular filtration rate estimated by CKD-EPI formula at months 3 and 6 then every 6 months
Change from baseline in proteinuria (g/d) or proteinuria /creatinuria (g/g) | From baseline and up to 36 months
  Change from baseline in proteinuria (g/d) or proteinuria /creatinuria (g/g) at months 3 and 6 then every 6 months
Proportion of patients who used at least one diuretic | Up to 36 months
Change from baseline in quality of life | From baseline and up to 36 months
  Change from baseline in quality of life assessed by PROMIS-29 survey each year

CONTACTS AND LOCATIONS:
Overall Officials: Bénédicte Sautenet, MD, Principal Investigator — University Hospital, Tours
Locations (40):
- France (40):
  - Department of Nephrology, University Hospital of Angers, Angers
  - Department of Nephrology, University Hospital of Bordeaux, Bordeaux
  - AUB Santé foundation, Brest, Brest
  - Department of Nephrology, University Hospital of Brest, Brest
  - Department of Nephrology, Hospital of Chalon-sur-Saône, Chalon-sur-Saône
  - Department of Nephrology, Hospital of Chartres, Chartres
  - Department of Nephrology, University Hospital of Clermont-Ferrand, Clermont-Ferrand
  - Department of Nephrology, Hospital of Colmar, Colmar
  - Department of Nephrology, University Hospital of Grenoble, Grenoble
  - Department of Nephrology, Hospital of Haguenau, Haguenau
  - Department of Nephrology, Departemental Hospital of Vendée, La Roche-sur-Yon
  - ECHO Santé Association, Le Mans, Le Mans
  - Department of Nephrology, Hospital of Le Puy en Velay, Le Puy-en-Velay
  - Department of Nephrology, University Hospital of Lille, Lille
  - Department of Nephrology, University Hospital of Limoges, Limoges
  - AUB Santé foundation, Lorient, Lorient
  - Department of Nephrology, University Hospital of Lyon, Lyon
  - Department of Nephrology, University Hospital of Marseille, Marseille
  - Department of Nephrology, Regional Hospital of Metz, Metz
  - Department of Nephrology, Régional Hospital of Mulhouse, Mulhouse
  - Department of Nephrology, University Hospital of Nantes, Nantes
  - ECHO Santé Association, Nantes, Nantes
  - Department of Nephrology, University Hospital of Nîmes, Nîmes
  - Department of Nephrology, Hospital of Orléans, Orléans
  - Department of Nephrology, European Hospital Georges Pompidou, AP-HP, Paris
  - Department of Nephrology, Necker Hospital, AP-HP, Paris
  - Department of Nephrology, Bichat Hospital, AP-HP, Paris
  - Department of Nephrology, Tenon Hospital, AP-HP, Paris
  - Department of Nephrology, Hospital of Perpignan, Perpignan
  - Department of Nephrology, University Hospital of Reims, Reims
  - Department of Nephrology, University Hospital of Rennes, Rennes
  - Department of Nephrology, Hospital of Roubaix, Roubaix
  - Department of Nephrology, University Hospital of Rouen, Rouen
  - Department of Nephrology, University Hospital of Saint Etienne, Saint-Etienne
  - ECHO Santé Association, Saint Herblain, Saint-Herblain
  - Department of Nephrology, Hospital of Saint Malo, St-Malo
  - Department of Nephrology, Hospital of Strasbourg, Strasbourg
  - Department of Nephrology, University Hospital of Tours, Tours
  - Department of Nephrology, Hospital of Valenciennes, Valenciennes
  - Department of Nephrology, University Hospital of Nancy, Vandœuvre-lès-Nancy